CLINICAL TRIAL: NCT06588205
Title: Multicenter, Observational, Retrospective-prospective Study Exploring the Clinical Impact of MYC Aberrations and Their Relationship With Microenvironment in Diffuse Large B Cell Lymphoma and High-Grade B Cell Lymphoma
Brief Title: Exploring the Clinical Impact of MYC Aberrations and Their Relationship With Microenvironment in Diffuse Large B Cell Lymphoma and High-Grade B Cell Lymphoma
Acronym: FIL_MIMYC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_MIMYC
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements
Keywords: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; MYC; BCL2; BCL6; Double Hit; Triple Hit; lymphoma micro-environment
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient affected by DLBCL or HGBL with MYC alterations treated with standard R-chemotherapy regimens as first line treatment

SUMMARY:
This is a observational, retrospective and prospective study designed to assess the potential correlations between MYC alterations, lymphoma mutational landscape and functional immune contextures in Diffuse Large B-cell Lymphoma or High-Grade B-cell Lymphoma

DETAILED DESCRIPTION:
Diffuse large B-cell lymphomas (DLBCL) and high-grade B-cell lymphomas (HGBCL) are a group of heterogeneous diseases representing more than a third of lymphomas in adults. 5-years overall survival of patients affected by DLBCL and HGBCL is around 70-60% and efficient prognostic markers are warranted to improve patients' survival by better tailored therapeutical approaches.

Genetic rearrangements of the MYC gene occur in 5-10% of DLBCL at diagnosis, and the presence of double translocations involving both MYC and BCL2 ("double-hit", DH), associated or not with BCL6 ("triple-hit", TH) translocation, is associated with unfavorable prognostic impact.

Intensification of treatment compared to standard chemotherapy (R-CHOP) appears to reduce the risk of recurrence in patients with DH or TH lymphomas, but a survival advantage has not been demonstrated.

Numerical changes in MYC (gain of copy number, GCN) may also affect the outcome of patients with DLBCL, but their prognostic relevance and the benefit of treatment intensification is still controversial.

Additionally, novel scientific evidence indicates a contribution of lymphoma micro-environment (LME) in disease genomic subtype and patient prognosis.

We aimed this study at investigating potential biological links between MYC aberrations, lymphoma mutational landscape and functional immune contextures in DLBCL and HGBCL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nodal and extranodal Diffuse Large B Cell Lymphoma, High Grade B Cell Lymphomas (including low-grade transformed lymphomas; double and triple hit; 11q aberration; not otherwise specified) after 1st January 2019
* Presence of one MYC translocation or gain of copies (GCN: > 3 copies in more than 30% of the nuclei) or amplification evaluated by FISH
* Availability of immunohistochemical analysis of CD10, Bcl6, MUM1, Bcl2, Myc, Ki67
* Have received curative treatment (e.g. R-CHOP, R DA EPOCH, intensified "Burkitt like" chemotherapies) as first-line therapy
* Histological material of adequate size and quality to perform histological review with any additional investigations (immunohistochemistry, FISH and other molecular analysis). A FFPE block must be provided for patient enrollment.
* Age between 18 and 79 years

Exclusion Criteria:

* Primary lymphomas of the central nervous system, plasmablastic lymphoma, Burkitt's lymphoma, primary mediastinal B lymphoma
* Have received palliative treatment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient affected by DLBCL or HGBL with MYC alterations treated with standard R-chemotherapy regimens as first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the histopathological, genetic, clinical characteristics and outcome of patients with DLBCL or HGBCL with MYC rearrangements or GCN (alone or in association with BCL2 and BCL6) treated with curative intent therapy | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Comparison of Progression Free Survival (PFS) according to genetic subgroups with or without intensified treatment

SECONDARY OUTCOMES:
Identify biological relationship between MYC aberration, gene mutations and patterns of immune microenvironment in B-cell lymphomas with DLBCL or high-grade morphology | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  % of patients with presence of MYC, BCL2 and/or BCL6 translocation evaluated by FISH
Identify biological relationship between MYC aberration, gene mutations and patterns of immune microenvironment in B-cell lymphomas with DLBCL or high-grade morphology | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  % of patients with presence of MYC gain of copy (GCN: > 3 copies in more than 30% of the nuclei) evaluated by FISH
Identify biological relationship between MYC aberration, gene mutations and patterns of immune microenvironment in B-cell lymphomas with DLBCL or high-grade morphology | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  % of patient with presence of MYC amplification evaluated by FISH
Identify putative prognostic and predictive biomarkers related to the lymphoma microenvironment | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Correlation between the microenvironment signature and patient Overall Survival (OS)
Analyze the impact of the type of therapy, standard or intensified (with or without autotransplantation), on the outcome in the different subgroups of patients | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Progression Free Survival comparison in the different subgroups of lymphomas and according to the type of treatment received
Assess the risk of central nervous system (CNS) recurrence and the impact of prophylaxis performed with intrathecal chemotherapy vs methotrexate intravenous | The endpoint will be evaluated from the beginning to the end of the study (up to 36 months)
  Progression Free Survival comparison in the different subgroups of lymphomas and according to the type of treatment received

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Lorenzi, MD, Principal Investigator — SC Anatomia Patologica - ASST Spedali Civili di Brescia
Locations (20):
- Italy (20):
  - A.O.U. SS. Antonio e Biagio e C. Arrigo - S.C.D.U. Ematologia, Alessandria
  - A.O.U. Ospedali Riuniti delle Marche - Clinica di Ematologia, Ancona
  - I.R.C.C.S. Istituto Tumori Giovanni Paolo II - U.O.C. Ematologia, Bari
  - ASST Spedali Civili - S.C. Ematologia, Brescia
  - I.R.C.C.S. Istituto di Candiolo - FPO, Candiolo
  - I.R.C.C.S. Istituto Oncologico Veneto - U.O.C. Oncoematologia, Castelfranco Veneto
  - ARNAS Garibaldi - U.O.C. Ematologia, Catania
  - A.S.T. Macerata - U.O.S.D Ematologia, Civitanova Marche
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda - S.C. Ematologia, Milan
  - Ospedale Maggiore Policlinico Fondazione IRCCS Ca' Granda - S.C. Ematologia, Milan
  - A.O.U. di Padova - U.O.C. Ematologia, Padua
  - I.R.C.C.S. Istituto Oncologico Veneto - U.O.C. Oncologia 1, Padua
  - AUSL Modena sede di Sassuolo - UOSD di Oncologia Area Sud, Sassuolo
  - U.O.C. Ematologia - A.O.U. Senese, Siena
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia U, Torino
  - ULSS 2 Ospedale Ca' Foncello - U.O.C. Ematologia, Treviso
  - A.O. Cardinale "G. Panico" - U.O.C Ematologia e Trapianto Midollo Osseo, Tricase
  - A.S.U. Giuliano Isontina - S.C. Ematologia, Trieste
  - A.O.U.I. di Verona - Ematologia, Verona

IPD SHARING:
Plan to Share IPD: Undecided